CLINICAL TRIAL: NCT03985215
Title: The Value of Follow-Up After Childhood Acute Lymphoblastic Leukaemia in Denmark - Family Perspectives
Status: Withdrawn | Type: Observational
Why Stopped: Overlapping with another danish questionnaire study
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-051-000001
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-07

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Surveys and Questionnaires
Keywords: Aftercare
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Pediatric Quality of Life Inventory questionnaire. Self-designed questionnaire.

SUMMARY:
The aim of the study is to evaluate the family perspective on follow-up programs after treatment for childhood acute lymphoblastic leukaemia. It is relevant when new follow-up programs are to be designed.

DETAILED DESCRIPTION:
More than 90 % of paediatric patients with acute lymphoblastic leukaemia (ALL), treated on the Nordic Society of Pediatric Hematology and Oncology (NOPHO) ALL-2008 protocol, are alive five years after diagnosis. The main reason for treatment failure being relapse.

The risk of relapse after treatment for ALL is highest within the first two years after cessation of maintenance therapy. Therefore, it has been routine in most countries to follow-up patients in the outpatient clinic every one or two months during the first years after end of therapy for ALL in order to detect recurrence and possible late sequelae at an early stage.

In children with ALL there are only a few studies on the value of routine follow-up, including haematological status after cessation of maintenance therapy. These studies showed that approximately 90% of the relapses were diagnosed in children with symptoms of leukaemia progression and that routine blood tests and clinical follow-ups were of little value. It is well known that there are other issues besides the risk of relapse, which are relevant for families after cessation of ALL therapy i.e. risk of late effects of treatment, psychosocial problems related to the child's return to "normal" life etc. These issues will also have an impact upon how the follow-up programs are planned. The investigators will study the family perspectives on follow-up during the first 5-years after cessation of maintenance therapy in a Danish cohort of children treated according to the NOPHO ALL-2008 protocol.

The investigators will conduct a cross-sectional study. Outcomes are patient-reported as the measurement instrument used is questionnaires. Eligible families are families with children diagnosed with acute lymphoblastic leukaemia in Denmark and being in the period 0-5 years after cessation of maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-precursor ALL and T-ALL enrolled in the NOPHO ALL-2008 trial
* Age group 1.0-14.9 years.
* Patients treated on one of the four Danish Paediatric oncology departments
* Patients in the time period 0-5 years after cessation of maintenance therapy for ALL

Exclusion Criteria:

* A history of recurrence or second malignancies
* Bone marrow transplantation
* Down syndrome
* If, due to language barriers, the family is unable to complete the questionnaire.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Questionnaires will be sent to all the possible families in Denmark with a child in the period of 0-5 years after cessation of maintenance therapy for ALL.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Degree of parental concern | A single point in time when questionnaires are answered. The specific time point being 0-5 years after end of ALL treatment.
  Self-designed questionnaire. Six items scored on a scale 1-7. Higher values represent a worse outcome. An average is calculated over the six items.
  An item evaluating the need for extra visits on a scale 1-3. Higher values represent a worse outcome.
  An item evaluating parental reported worries about the future on a scale 1-5. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Satisfaction with the follow-up program | A single point in time when questionnaires are answered. The specific time point being 0-5 years after end of ALL treatment.
  Self-designed questionnaire. An item evaluating satisfaction the time interval between visits on a scale 1-3. Higher values represent a worse outcome.
PedsQL scores | A single point in time when questionnaires are answered. The specific time point being 0-5 years after end of ALL treatment.
  Pediatric Quality of Life Inventory questionnaire (the parent proxy). A validated measure of health-related quality of life.
The amount of self-reported side effects | A single point in time when questionnaires are answered. The specific time point being 0-5 years after end of ALL treatment.
  Self-designed questionnaire. Fifteen items scored on a scale 1-7. Higher values represent a worse outcome. An average is calculated over the fifteen items.
  An item evaluating the duration of the time period before the child was able to attend day-care/school on a scale 1-5. Higher values represent a worse outcome.
Strategy of the families between follow-up visits | A single point in time when questionnaires are answered. The specific time point being 0-5 years after end of ALL treatment.
  Self-designed questionnaire. In need of advice between visits what are the strategy of the participants: seeking hospital, general practitioner or postponing till next scheduled visit.

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Jensen, MD, Principal Investigator — Aarhus Universitet
Locations (1):
- Karen Schow Jensen, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No